CLINICAL TRIAL: NCT04926064
Title: Young Children's Sleep Patterns and Problems Among Turkish Children: Cross-sectional Study From a Nationally Representative Sample
Brief Title: Young Children's Sleep Patterns and Problems Among Turkish Children
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Perran Boran, Professor of Pediatrics, Marmara University
Other Study IDs: 09.2021.489
Record Dates: First submitted 2021-06-08; First posted 2021-06-14 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2022-08

CONDITIONS: Child Behavior Problem
Keywords: sleep; insomnia; children
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sleep is important for optimal child growth, development, and family functioning. Behavioral pediatric insomnia is one of the most prevalent sleep disorders identified in young children. Well-child visits represent an important setting for addressing concerns regarding the child's sleep patterns and sleep problems.

Investigators aimed to describe sleep/wake patterns of young children, evaluate the associations between parental depressive, and anxiety symptoms, parental involvement in child-care, sleep-related behaviors and children's sleep parameters.

The study has a descriptive cross-sectional study design. An estimated sample size was 2089 participants considering the number of children aged between 6-36 months in the country, and the estimated prevalence of Behavioral Insomnia being 30%. A multi-stage stratification is used to calculate the number of participants to be taken at the level of 12 geographical regions according to Nomenclature of Territorial Units for Statistics (NUTS-1). A sleep study group is established by the study coordinator, and researchers running a well-child outpatient clinic from each region across the country are included.

Investigators invite mothers of children aged 6 to 36 months who either visited for a well-child outpatient clinic or in the waiting list for follow up to complete the online questionnaire about their children's sleep/wake patterns utilizing mailing lists obtained from the outpatient clinics. Recruitment will take place from April to June 2021. The questionnaire included Brief Infant Sleep Questionnaire (BISQ), Edinburgh Postnatal Depression Scale (EPDS) and Generalized Anxiety Disorder (GAD-7) scale, and separate questions on fathers' involvement in child care, and sociodemographic characteristics. An online google survey is developed on the google platform securing data collection by a confidential log in system which can be filled out from smartphones, tablet or computer. The questionnaire takes approximately 20 minutes to complete.

DETAILED DESCRIPTION:
Sleep is important for optimal child growth, development, and family functioning. Behavioral pediatric insomnia is one of the most prevalent sleep disorders identified in young children. Well-child visits represent an important setting for addressing concerns regarding the child's sleep patterns and sleep problems.

Investigators aimed to describe sleep/wake patterns of young children, evaluate the associations between parental depressive, and anxiety symptoms, parental involvement in child-care, sleep-related behaviors and children's sleep parameters.

The study has a descriptive cross-sectional study design. According to the formula for the known number of individuals in the universe [Sample formula with known number of individuals n = [Np(1-p)]/ [(d2/Z21-α/2*(N-1)+p*(1-p)], (α=0.05, p=0.32, d=0.02) the sample size to represent the population was found to be 2089, considering the number of children aged between 6-36 months in the country, and the estimated prevalence of Behavioral Insomnia being 30%. A multi-stage stratification is used to calculate the number of participants to be taken at the level of 12 geographical regions according to Nomenclature of Territorial Units for Statistics (NUTS-1). A sleep study group is established by the study coordinator, and researchers running a well-child outpatient clinic from each region across the country are included.

Investigators invite mothers of children aged 6 to 36 months who either visited for a well-child outpatient clinic or in the waiting list for follow up to complete the online questionnaire about their children's sleep/wake patterns utilizing mailing lists obtained from the outpatient clinics. Recruitment will take place from April to June 2021. The questionnaire included Brief Infant Sleep Questionnaire (BISQ), Edinburgh Postnatal Depression Scale (EPDS) and Generalized Anxiety Disorder (GAD-7) scale, and separate questions on fathers' involvement in child care, and sociodemographic characteristics. An online google survey is developed on the google platform securing data collection by a confidential log in system which can be filled out from smartphones, tablet or computer. The questionnaire takes approximately 20 minutes to complete.

ELIGIBILITY:
Inclusion Criteria:

* mothers of healthy infants aged between 6 to 36 months

Exclusion Criteria:

infants <37 gestational week, congenital disease, neurodevelopmental disorder, use of drugs that can affect sleep such as diphenhydramine, Obstructive Sleep Apnea diagnosis

Ages: 6 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: mothers of healthy infants aged between 6 to 36 months
Sampling Method: Probability Sample
Enrollment: 2434 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-08-14 (Actual)

PRIMARY OUTCOMES:
Sleep wake patterns | Baseline
  Sleep wake patterns of children aged between 6-36 months
Sleep problem | Baseline
  Maternal report of sleep problem

SECONDARY OUTCOMES:
maternal depression | Baseline
  maternal depression score assessed with Edinburgh Postnatal Depression Scale
maternal anxiety | baseline
  maternal anxiety score assessed with Generalized Anxiety Scale-7
paternal involvement in child care | baseline
  paternal involvement will be assessed with 5 questions

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Turkey (Türkiye)